CLINICAL TRIAL: NCT01055210
Title: Optimisation of Cardiac Resynchronisation Therapy by Non-invasive Cardiac Output - The CHOICE2 Study
Acronym: CHOICE2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Dundee (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ELD002
Record Dates: First submitted 2010-01-22; First posted 2010-01-25 (Estimated); Last update posted 2018-12-03 (Actual); Status verified 2010-01

CONDITIONS: Heart Failure; Cardiac Resynchronisation Pacemakers
Keywords: Heart Failure; Pacemakers
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Optimisation of VV delay — Programmed VV delay altered on device

SUMMARY:
An evaluation of the role of resting and exercise cardiac output measurement, by the inert gas rebreathing method, in optimisation of patients with cardiac resynchronisation pacemakers.

ELIGIBILITY:
Inclusion Criteria:

* Cardiac Resynchronization Device in situ for Heart Failure

Exclusion Criteria:

* Unable to cope with mouthpiece
* Estimated life expectancy < 6 months

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2010-02; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
6 minute hall walk test | 4 months

SECONDARY OUTCOMES:
Echocardiographic measures of desynchrony | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Anna- Maria Choy, Principal Investigator — University of Dundee
Locations (1):
- University of Dundee, Dundee, United Kingdom